CLINICAL TRIAL: NCT02775279
Title: Short Telomere Length in Peripheral Blood Leukocyte Predicts the Risk of Acute Coronary Syndrome
Brief Title: Association Between Telomere Length and Risk of Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Wenyi Guo, Professor of Department of Cardiovascular Medicine, Air Force Military Medical University, China
Other Study IDs: XJ20160520
Record Dates: First submitted 2016-05-14; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome, telomere length, predictive factor
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Telomeres consist of a tandem TTAGG repeat located at ends of linear chromosomes of eukaryote cells that often decrease in length over time (largely due to oxidative damage and the end replication problem during cell division) and may trigger cellular senescence once telomere become critically short
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute coronary syndrome group: 200 consecutive patients were recruited, who have diagnosed with acute coronary syndrom(ACS) by quantitative coronary angiography.
- Control group: The 200 healthy controls without previous CHD history were recruited from individuals who visited investigator's hospital for physical examination during the same time period as the case enrollment.

SUMMARY:
Compelling epidemiological evidence indicates that alterations length of telomere, are associated with the initiation and development of ischemic heart disease. This study was undertaken to investigate whether mtDNA copy number in peripheral blood leukocyte could be used as a risk predictor for acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

-1.History of documented myocardial infarction; 2.Prior coronary revascularization intervention (coronary artery bypass graft surgery or percutaneous coronary intervention); 3.The presence of≥50% stenosis in one or more coronary arteries identified during cardiac catheterization;

Exclusion Criteria:

-1.History of malignancy or end-stage renal disease; 2.Blood transfusion within one month or prior bone marrow transplantation 3.Patients who reluctant to sign informed consent

Ages: 18 Years to 85 Years | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 200 eligible ACS patients were anticipated to include in this study.Moreover, The 200 healthy controls without previous CHD history were also recruited from individuals who visited investigator's hospital for physical examination during the same time period.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Relative telomere length | From date of percutaneous coronary intervention until the date of discharging from hospital, assessed up to 5 days
  the ratio of telomere repeat copy number(T) to the hemoglobin(HGB) copy number (S) was determined for each sample using standard curves. The derived T/S ratio was proportional to the relative telomere length(RTL). In the second step, the T/S ratio of each sample was normalized to a calibrator DNA to standardize between different PCR runs. The calibrated T/S ratio was then used as the measurement of RTL in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No